CLINICAL TRIAL: NCT07046962
Title: Comparison of Macronutrient Content of Breast Milk Collected From Mothers Using Three Different Milking Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Macronutrient
Record Dates: First submitted 2025-05-22; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breastmilk; Breastmilk Expression; Breastmilk Collection; Human Milk/Breastfeeding; Macronutrients
Keywords: Anne sütü,; macrobesin,; protein,; yağ,; karbonhidrat
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Type Device: hand expressing breast milk (Experimental): Samples were taken by hand milking the mother's milk.
  Interventions: Other: Intervention Type Device: Hand pumping breast milk
- Intervention Type Device: breast milk expression group with manual pump (Experimental): Breast milk was obtained with a manual pump.
  Interventions: Other: Intervention Type Device: Manual pump expressing breast milk
- Intervention Type Device: expressing breast milk with electric pump (Experimental): Breast milk was expressed with an electric pump.
  Interventions: Other: Intervention Type Device: Electric pumping breast milk

INTERVENTIONS:
Other: Intervention Type Device: Manual pump expressing breast milk — Since this study aimed to examine the macronutrient content of milks expressed from the same mother with three different methods, one day apart, the data collection process was carried out in stages. The methods determined by randomization were hand expressing breast milk, hand pumping and electric pumping.
  Hand expressing: Milk was expressed by hand until the milk flow stopped at the mother's breast. While the baby was sucking from one breast, the other breast was milked, and a 10 cc sample was taken from the collected milk and placed in sterile fallopian tubes.
  Arms: Intervention Type Device: breast milk expression group with manual pump
Other: Intervention Type Device: Hand pumping breast milk — Since this study aimed to examine the macronutrient content of milk expressed from the same mother with three different methods, one day apart, the data collection process was carried out in stages. The methods determined by randomization were hand expressing breast milk, manual pump expressing and electric pump expressing.
  Manual pump expressing: Milk was expressed with a manual pump until the milk flow stopped in the mother's breast. While the baby was sucking from one breast, the other breast was milked, and a 10 cc sample was taken from the collected milk and placed in sterile fallopian tubes.
  Arms: Intervention Type Device: hand expressing breast milk
Other: Intervention Type Device: Electric pumping breast milk — Since this study aimed to examine the macronutrient content of milk expressed from the same mother with three different methods, one day apart, the data collection process was carried out in stages. The methods determined by randomization were hand expressing breast milk, manual pump expressing and electric pump expressing.
  Electric pump expressing: Milk was expressed with an electric pump until the milk flow stopped in the mother's breast. While the baby was sucking from one breast, the other breast was milked, and a 10 cc sample was taken from the collected milk and placed in sterile fallopian tubes.
  Arms: Intervention Type Device: expressing breast milk with electric pump

SUMMARY:
The aim of this study is to compare the macronutrient content of mature milk obtained from mothers using three different methods: hand milking, manual pumping and electric machine. This study, which was conducted with an experimental design, included 31 mothers who met the sample criteria. The macronutrient content of mature milk obtained from mothers with term babies using three different milking methods was examined by providing the highest level of standardization in the sample. A nutrition plan was applied to the mothers three days before milk samples were taken and on the milking days. Milk was milked from the mothers according to the three different methods specified in the randomization one day apart. Data were obtained with the Introductory Information Form, Breast Milk Information Form, Breast Milk Follow-up Form and Daily Food Consumption Record Form. Frozen milk samples were analyzed with Miris® HMATM to determine protein, fat, carbohydrate and energy values. Data were analyzed using the R programming language version 4.4.1.

DETAILED DESCRIPTION:
The World Health Organization (WHO) and the United Nations International Children's Emergency Fund (UNICEF) recommend that breastfeeding should be initiated within half an hour postpartum, that the baby be given only breast milk for the first six months, and that breastfeeding should be continued until the age of two and beyond with the addition of appropriate complementary foods after six months. Breast milk, a unique food, is a complex biological system with macronutrients, micronutrients, and bioactive factors. The content of breast milk varies among mothers, as well as depending on the gestational week, postnatal age, lactation period, time of day, and from the beginning to the end of breastfeeding. In this dynamic process, the content is adjusted according to the baby's needs. The most ideal way to give breast milk to the baby is for the baby to suckle. The most appropriate form of nutrition for babies is first to be breastfed by their own mother, followed by the artificial feeding of their own mother's expressed milk, donor breast milk, and finally formula. Due to some factors related to the baby and the mother, it may be necessary to express milk instead of breastfeeding directly. If the mother and baby cannot meet after birth, it is recommended to express milk within the first six hours and give breast milk to the baby. In expressing breast milk, hand expression or pumping (electric pump and manual pump) methods are used. In the review published in Cochrane in 2016, no recommendation was made as to which method is superior, and it was reported that there were differences in terms of participants, interventions and outcome variables in the studies conducted. In the Healthy Term Baby Feeding Guide of the Turkish Neonatology Association (2024), it is stated that every mother should be taught how to express milk before discharge, and especially mothers who cannot breastfeed their babies should be trained on expressing milk from the first hour. Although it is stated in this guide that milk expression methods are not superior to each other as long as they are done appropriately; It is reported that the most appropriate milking method varies according to when and why the milking will be done after birth and the individual characteristics of the mother/baby duo, that simple and inexpensive methods such as hand milking, massage and warming the breasts can be as effective as or even more effective than electric pumps, and that there is still a need for studies with a high level of evidence to show which method is superior. When the studies conducted in the literature to determine the effect of the milk expression method on the content of breast milk were evaluated, it was seen that there was no standardization and some important deficiencies. In a systematic review conducted in 2021, the effect of the breast milk expression method on milk content was examined. In the study, studies conducted up to May 30, 2021 in six databases (Pubmed, Web of Science, MEDLINE, Science Direct, CINAHL and Cochrane) were examined, 258 studies were reached as a result of the screening, and six studies on the subject were evaluated. As a result of the study; It has been stated that the protein and carbohydrate content in breast milk does not change according to the milking method, but the fat content is affected by the milking method. In this study, it has been reported that there is no standardization of the variables affecting the breast milk content in the studies conducted in the literature, and that there is a need for studies in which all variables are standardized. When the studies conducted in the literature on the subject of the study were evaluated, it was seen that: content analysis was performed on colostrum, transitional milk or mature milk, but the foremilk or hindmilk was not clearly specified, the lactation stage of the mother was not specified, the breast from which the milk was examined, the time of day it was taken was not specified, there was no information on the mother's breast being accustomed to milking, the expression duration was not specified during machine or manual expression , the lack of information on how to adjust the machine modes during machine expression, how long after the last breastfeeding the milk was examined, the nutritional status of the mother, BMI, the gender of the baby, whether the baby is exclusively breastfed, gestational week of the infant, and exclusion of variables affecting the macronutrient content of breast milk. In the comprehensive literature review, it was concluded that studies were not conducted on sufficiently standardized samples in terms of basic variables affecting breast milk content. It was stated that there were methodological limitations in the studies conducted to examine the content of breast milk collected by different methods in terms of macronutrients, the variables that may cause the content to change were not sufficiently taken into account in the studies, and there is a need for standardization studies.

ELIGIBILITY:
Inclusion Criteria:

* The Inclusion Criteria for Mothers in the Study Sample;
* The mother must be primigravida
* The mother must have given birth normally
* The mother must be breastfeeding her baby only
* The mother must not have a diagnosed health problem related to nutrition
* The mother must be open to communication and cooperation
* The mother must volunteer to participate in the study
* The mother must be at least literate
* The mother must be over the age of 18
* The mother must not be a vegetarian
* The mother must not smoke
* The mother must not have a diagnosed breast trauma (mastitis, abscess, etc.) - The mother must not use any herbal tea or medication other than the doctor's recommendation
* The mother's body mass index must be within normal values (18.5 to 24.9) before pregnancy (WHO, 2015).

The mother must not be an immigrant/refugee/asylum seeker - The mother must have a smartphone and internet access

Exclusion Criteria:

* Exclusion Criteria for Mothers:
* The mother wants to leave the study
* The mother has a sudden trauma/health problem that prevents her from participating in the study
* The mother has moved to another city
* The mother has an anatomical condition that prevents breastfeeding in both breasts (absence of breast, burn, loss of breast tissue, etc.)
* The mother is an athlete

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast milk samples were taken from lactating mothers.
Enrollment: 31 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Protein content of mature breast milk measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The macronutrient content of the mature breast milk-including protein (g/100 mL) was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form.
  Unit of Measure:
  Protein (g/100 mL)
Energy content of mature breast milk measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The energy content of the mature breast milk-including energy (kcal/100 mL)-was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk energy content (kcal/100 mL).
Fat content of mature breast milk measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The fat content of the mature breast milk-fat (g/100 mL) was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk Fat (g/100 mL).
Carbohydrate content of mature breast milk measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Breast milk samples collected from each mother (10 mL) were stored at -18 °C and later thawed by a Nutrition and Dietetics researcher at 0-4 °C within 24 hours in the Nutrition and Dietetics Department Laboratory. To ensure reliability, each milk sample was analyzed twice. The carbohydrate of the mature breast milk-including carbohydrate (g/100 mL), was determined using the Miris® Human Milk Analyzer™ (Miris AB, Uppsala, Sweden). The analysis results were recorded in the Breast Milk Tracking Form. "Breast milk carbohydrate content (g/100 mL), measured using Miris® Human Milk Analyzer Unit of Measure

SECONDARY OUTCOMES:
Comparison of energy content of breast milk by expression method (hand, manual pump, electric pump), measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Mature breast milk samples (10 mL) were collected from lactating mothers between postpartum days 2 and 23 using three different expression methods: hand expression, manual breast pump, and electric breast pump. Each method was used for a separate milk collection. All samples were stored at -18 °C, then thawed at 0-4 °C and analyzed within 1 month. Energy content (kcal/100 mL) was measured using the Miris® Human Milk Analyzer™. Results were recorded in the Breast Milk Tracking Form. Comparisons will be made between the three expression method groups to assess differences in milk composition.
  Energy (kcal/100 mL)
  Differences in breast milk energy content among expression methods will be analyzed using appropriate statistical tests (e.g., repeated measures ANOVA or Kruskal-Wallis test, depending on distribution).
Comparison of protein content of breast milk by expression method (hand, manual pump, electric pump), measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Mature breast milk samples (10 mL) were collected from lactating mothers between postpartum days 2 and 23 using three different expression methods: hand expression, manual breast pump, and electric breast pump. Each method was used for a separate milk collection. All samples were stored at -18 °C, then thawed at 0-4 °C and analyzed within 1 month. protein content (g/100 mL) was measured using the Miris® Human Milk Analyzer™. Results were recorded in the Breast Milk Tracking Form. Comparisons will be made between the three expression method groups to assess differences in milk composition.
  Protein (g/100 mL)
  Differences in breast milk protein content among expression methods will be analyzed using appropriate statistical tests (e.g., repeated measures ANOVA or Kruskal-Wallis test, depending on distribution).
Comparison of fat content of breast milk by expression method (hand, manual pump, electric pump), measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Mature breast milk samples (10 mL) were collected from lactating mothers between postpartum days 2 and 23 using three different expression methods: hand expression, manual breast pump, and electric breast pump. Each method was used for a separate milk collection. All samples were stored at -18 °C, then thawed at 0-4 °C and analyzed within 1 month. Fat content (g/100 mL) was measured using the Miris® Human Milk Analyzer™. Results were recorded in the Breast Milk Tracking Form. Comparisons will be made between the three expression method groups to assess differences in milk composition.
  Fat (g/100 mL)
  Differences in breast milk fat content among expression methods will be analyzed using appropriate statistical tests (e.g., repeated measures ANOVA or Kruskal-Wallis test, depending on distribution).
Comparison of Carbohydrate content of breast milk by expression method (hand, manual pump, electric pump), measured by Miris® Human Milk Analyzer™ | Three consecutive postpartum days (Days 23-25)
  Mature breast milk samples (10 mL) were collected from lactating mothers between postpartum days 2 and 23 using three different expression methods: hand expression, manual breast pump, and electric breast pump. Each method was used for a separate milk collection. All samples were stored at -18 °C, then thawed at 0-4 °C and analyzed within 1 month. Carbohydrate (g/100 mL) content was measured using the Miris® Human Milk Analyzer™. Results were recorded in the Breast Milk Tracking Form. Comparisons will be made between the three expression method groups to assess differences in milk composition.
  Carbohydrate (g/100 mL)
  Differences in breast milk Carbohydrate content among expression methods will be analyzed using appropriate statistical tests (e.g., repeated measures ANOVA or Kruskal-Wallis test, depending on distribution).

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Karataş, Professor, Study Director — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The article will be shared after publication.